CLINICAL TRIAL: NCT02829775
Title: Extension Protocol for Patients With Chronic Myelogenous Leukemia, Malignant Melanoma or Renal Cell Carcinoma That Have Responded to Treatment With Pegylated-Interferon α-2a or Roferon-A® in Prior Clinical Studies
Brief Title: A Study of Continued Treatment Among Participants Who Have Responded to Peginterferon Alfa-2a (Pegasys®) or Recombinant Interferon Alfa-2a (Roferon-A®) in Prior Clinical Studies
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NO17754; 2004-002093-30 (EudraCT Number)
Record Dates: First submitted 2016-07-06; First posted 2016-07-12 (Estimated); Results first posted 2016-11-17 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Myelogenous Leukemia; Malignant Melanoma; Renal Cell Carcinoma
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Melanoma; Carcinoma, Renal Cell | interventions — peginterferon alfa-2a; Interferon alpha-2

ARMS (1):
- Interferon Alfa-2A in Cancer Participants (Experimental): Participants who responded to interferon alfa-2A (either pegylated interferon alfa-2A or recombinant interferon alfa 2A) treatment during the parent study will continue to receive the same treatment in this study. Pegylated interferon alfa-2A will be administered subcutaneously once weekly and recombinant interferon alfa 2A will be administered subcutaneously once daily, until disease progression, withdrawal, or death whichever occurs first (up to approximately 3 years).
  Interventions: Drug: Pegylated Interferon Alfa-2a; Drug: Recombinant Interferon Alfa 2a

INTERVENTIONS:
Drug: Pegylated Interferon Alfa-2a — Participants will maintain the same dose they were receiving in the parent protocol.
  Other Names: Pegasys
Drug: Recombinant Interferon Alfa 2a — Participants will maintain the same dose they were receiving in the parent protocol.
  Other Names: Roferon-A

SUMMARY:
This open label extension study will give an opportunity to the participants that have responded to the treatment with Pegylated-Interferon Alfa-2a (Pegasys) or Recombinant Interferon Alfa-2a (Roferon-A®) in prior clinical studies NO15753 (NCT00003542) for Renal Cell Carcinoma (RCC), NO15764 (NCT number not available) and NO16006 (NCT02736721) for Chronic Myelogenous Leukemia (CML), and NO16007 (NCT number not available) for Malignant Melanoma (MM).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have completed protocol NO15753, NO15764, NO16006 or NO16007 and responded to treatment at the end of the trial as defined in the parent protocol
* CML participants must have a confirmed cytogenetic complete response within 2 months of entering the extension study. MM and RCC participants must have tumour assessments verifying stable or better response within 2 months of entering the extension study

Exclusion Criteria:

* Pregnant or lactating women
* Refusal to use adequate contraceptive measures among men and women of childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (7):
- Sofia, Bulgaria
- Halifax, Nova Scotia, Canada
- Lucknow, India
- Moscow, Russia
- Košice, Slovakia
- Durban, South Africa
- Valencia, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 9 participants were recruited in the study: 8 participants from study NO16006 (NCT02736721) and 1 participant from study NO16007 (NCT number not available).
Groups:
- Interferon Alfa-2A in Cancer Participants: Participants who responded to interferon alfa-2A (either pegylated interferon alfa-2A or recombinant interferon alfa 2A) treatment during the parent study continued to receive the same treatment in this study. Pegylated interferon alfa-2A was administered subcutaneously once weekly and recombinant interferon alfa 2A was administered subcutaneously once daily, until disease progression, withdrawal, or death whichever occurred first (up to approximately 3 years).
Period: Overall Study
Arm/Group | Interferon Alfa-2A in Cancer Participants
Started | 9
Completed | 4
Not Completed | 5
Not completed — Death | 1
Not completed — Withdrawal by Subject | 3
Not completed — Disease remission | 1

BASELINE CHARACTERISTICS:
Population: All participants who were recruited in the study.
Arm/Group | Interferon Alfa-2A in Cancer Participants
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (18.3)
Gender [Count of Participants; unit: Participants]
  Female | 2
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship to the study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; Initial or prolonged inpatient hospitalization; Life-threatening experience (immediate risk of dying); Persistent or significant disability or incapacity; and congenital anomaly.
Time Frame: Baseline up to approximately 3 years
Population: All participants who were recruited in the study.
Measure: Number; unit: participants
Arm/Group | Interferon Alfa-2A in Cancer Participants
Number analyzed (Participants) | 9
participants | 1

2. Secondary Outcome: Number of Participants With Overall Tumor Response
Description: Tumor response was assessed every 6 months using hematological evaluation or any other appropriate diagnostic techniques, as per standard of care practice. The complete response (CR) and partial response (PR) status were recorded from case report form.
Time Frame: Baseline until disease progression, withdrawal or death, whichever occurred earlier (assessed every 6 months up to approximately 3 years)
Population: All participants who were recruited in the study.
Measure: Number; unit: participants
Groups:
- Interferon Alfa-2A in Cancer Participants: Participants who responded to interferon alfa-2A (either pegylated interferon alfa-2A or recombinant interferon alfa 2A) treatment during the parent study will continue to receive the same treatment in this study. Pegylated interferon alfa-2A will be administered subcutaneously once weekly and recombinant interferon alfa 2A will be administered subcutaneously once daily, until disease progression, withdrawal, or death whichever occurred first (up to approximately 3 years).
Arm/Group | Interferon Alfa-2A in Cancer Participants
Number analyzed (Participants) | 9
participants
  CR | 9
  PR | 0

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 3 years
Description: All participants who were recruited in the study. Only SAEs were planned to be monitored during this extension study.
Arm/Group | Interferon Alfa-2A in Cancer Participants
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon Alfa-2A in Cancer Participants (N=9)
Lung Infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.